CLINICAL TRIAL: NCT06808243
Title: Modified Vascularized Interpostional Periosteal Connective Tissue Graft Versus Xenogeneic Collagen Matrix for Soft Tissue Augmentation Around Implant in Esthetic Zone (Comparative Study)
Brief Title: Modified Periosteal Tissue Graft vs Collagen Matrix for Soft Tissue Augmentation Around Implants: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, heba ahmed abdelmaged, Teaching assistant, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 543/84/2021; clinical trial (Registry Identifier: Minia University)
Record Dates: First submitted 2025-01-15; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Dental; Implant
Keywords: implant; connective tissue graft; xenogenic membrane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- modified vestibular interpositional periosteal connective tissue graft (Experimental): 10 patients received pedicled CTG (mVIP-CTG)
  Interventions: Procedure: connective tissue graft
- Xenogenic Collagen Membrane (Experimental): 10 patients received xenogenic collagen membrane
  Interventions: Device: xenogenic collagen membrane

INTERVENTIONS:
Procedure: connective tissue graft — 10 patients received mVIP-CTG
  Arms: modified vestibular interpositional periosteal connective tissue graft
Device: xenogenic collagen membrane — 10 patients received XCM
  Arms: Xenogenic Collagen Membrane

SUMMARY:
This clinical trial aims to evaluate the effectiveness of the Modified Vascularized Interpositional Periosteal Connective Tissue Graft (mVIP-CTG) compared to Xenogeneic Collagen Matrix (XCM) around immediate implant in esthetic zone . This study will assess outcomes such as keratinized tissue thickness, keratinized tissue width, pink esthetic score and radiographic buccal cortex thickness over a defined follow-up period. By comparing mVIP-CTG to XCM, the study seeks to determine which method provides superior clinical and aesthetic results for best soft tissue augmentation

DETAILED DESCRIPTION:
This study investigates two surgical techniques for managing peri-implant soft tissue deficiencies: the Modified Vascularized Interpositional Periosteal Connective Tissue Graft (VIP-CTG) and the Xenogeneic Collagen Matrix (XCM). Peri-implant soft tissue deficiencies, characterized by inadequate tissue volume or recession around dental implants, can lead to complications such as implant exposure, sensitivity, and aesthetic concerns. Conventional treatment methods aim to enhance soft tissue volume and improve the aesthetic and functional outcomes of implants.

The mVIP-CTG approach utilizes autogenous pedicle grafts to improve tissue thickness and width, potentially enhancing soft tissue integration and thickness around immediate implants. In contrast, XCM is a xenogenic membrane offering a minimally invasive alternative substitute for soft tissue regeneration.

The study design includes randomized assignment of participants to either the mVIP-CTG group or XCM group, with standardized surgical and follow-up protocols. Primary and secondary outcomes will include peri-implant soft tissue thickness, keratinized tissue width, pink esthetic score, and radiographic buccaal cortex thickness. Statistical analysis will evaluate the comparative effectiveness of both techniques in promoting peri-implant soft tissue regeneration and aesthetic recovery.

ELIGIBILITY:
Inclusion Criteria: -

* systemically healthy
* teeth indicated for extraction due to trauma or root fracture
* periodontally healthy
* Good oral health
* Selected patients of both sexes are 20-40 years old.

Exclusion Criteria:

* parafunctional habits
* smoking, alcoholism
* pregnancy
* lactation
* untreated periodontal diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
keratinized tissue thickness | baseline, 3 months, 6 months
  measurement of Kertinized tissue thickness around implant using endodontic file
keratinized tissue width | baseline, 3 months and 6 months
  measurement of keratinized tissue width using graduated UNC-15 Probe
buccal cortex thickness | baseline and 6 months
  measurement of buccal cortex thickness using CBCT

SECONDARY OUTCOMES:
pink esthetic score | baseline and 6 months
  measurement of pink aesthetic using visual scale of pink asethetic score

CONTACTS AND LOCATIONS:
Overall Officials: Heba Ah Abdel-maged, MSc, Principal Investigator — Minia University
Locations (1):
- Hospital of faculty of dentistry, Minia university, Minya, Egypt

DOCUMENTS (2):
  • Study Protocol (2021-11-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT06808243/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT06808243/SAP_001.pdf